CLINICAL TRIAL: NCT05872451
Title: The Difference in the Current Intensity for the Obturator Nerve Block According to the Presence or Absence of Neuromuscular Blockage
Brief Title: Current Intensity for the Obturator Nerve Block
Acronym: Current_ONB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chosun University Hospital (Other)
Responsible Party: Principal Investigator, Ki Tae Jung, Professor, Chosun University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ONB
Record Dates: First submitted 2023-05-12; First posted 2023-05-24 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Bladder Tumor
Keywords: Transurethral Resection of Bladder; Obturator Nerve; Nerve Block; Neuromuscular Blockade; Anesthesia, General
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Rocuronium

STUDY DESIGN:
Intervention Model Description: Patients undergoing TURP procedure under general anesthesia
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Current intensity (Experimental): 1. An I-gel mask is inserted for the mechanical ventilator of the patient who is sedated with propofol.
  2. For the ultrasound-guided obturator nerve (ON) block, and needle tip gradually advanced to the anterior branch of the ON. The current intensity for the stimulation of ON starts at 1.0 mA (using the sequential electrical nerve stimulation mode), and the needle is advanced gradually to the location where the contraction of the adductor longus muscle (ALM) occurs at 0.3-0.5 mA.
  3. After fixing the needle in that position, measure the current intensity.
  4. Then, rocuronium (0.6 mg/kg) is administered under quantitative neuromuscular-blockade monitoring.
  5. When the train-of-four count becomes 0, the current intensity is increased until the contraction of the ALM occurs.
  6. The current intensity is measured when the contraction of the ALM occurs.
  Interventions: Drug: Rocuronium Bromide; Diagnostic Test: Nerve stimulator

INTERVENTIONS:
Drug: Rocuronium Bromide — After measuring the initial current intensity, quantitative neuromuscular blockade monitoring is applied, and rocuronium (0.6 mg/kg) is administered.
  Other Names: Rocuronium
Diagnostic Test: Nerve stimulator — Measuring the minimum current intensity for the stimulation of the obturator nerve to show the contraction of the adductor longus muscle.
  Other Names: Stimuplex

SUMMARY:
The purpose of the present study was to find out the difference in current intensity required for nerve stimulation according to the presence or absence of neuromuscular blockade during the obturator nerve block procedure for TURP.

DETAILED DESCRIPTION:
During the transurethral resection of bladder tumors (TURBT) procedure under spinal anesthesia, the obturator nerve block is required to prevent the accidental movement of adductor longus muscles by electrical stimulation. However, during general anesthesia, the contraction of the adductor longus muscle would be lost due to deep neuromuscular blockade. However, some reports showed that the contraction of the adductor longus muscle occurs even in the deep neuromuscular blockade.

The current intensity for the nerve stimulation during nerve block is 0.3--0.5 mA when the needle tip is near the nerve. However, it is still unknown what current intensity is required to show the contraction of the adductor longus muscle when the patient is in a deep neuromuscular blockade.

Therefore, in this study, investigators aimed to determine the difference in current intensity required for nerve stimulation according to the presence or absence of neuromuscular blockade during obturator nerve block for TURP. In addition, investigators aimed to determine that the obturator nerve block is required during the TURP procedure in patients with deep neuromuscular blockade during general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing TURP procedure

Exclusion Criteria:

* Patients with anatomical or functional anomaly in the upper airways
* Patients with neuromuscular disease
* Patients with hip joint disorders
* BMI of < 18.5 or > 30.0 kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Initial current intensity | About 5 minutes after starting obturator nerve block procedure
  The current intensity for the stimulation of the obturator nerve starts at 1.0 mA (using the sequential electrical nerve stimulation mode), and the needle is advanced gradually to the location where the stimulus response occurs at 0.3-0.5 mA. After fixing the needle position in a position where contraction of the adductor longus muscle responds to the minimum current intensity, measure the current intensity.
Final current intensity | About 10 minutes after starting obturator nerve block procedure
  After administration of rocuronium (0.6 mg/kg), when the train-of-four count becomes 0, the current intensity for the stimulation of the obturator nerve is increased until the contraction of the adductor longus muscle occurs. The current intensity is measured when the contraction of the adductor longus muscle occurs.

SECONDARY OUTCOMES:
Current intensity after the administration of rocuronium (0.6 mg/kg) | Between 5 minutes and 10 minutes after starting obturator nerve block procedure
  After administration of rocuronium (0.6 mg/kg), the quantitative neuromuscular blockade monitoring using train-of-four is observed with 12 seconds interval. At each time point, the current intensity for the obturator nerve is increased until the contraction of the adductor longus muscle occurs. The current intensity at each time point is measured.

CONTACTS AND LOCATIONS:
Overall Officials: Ki Tae Jung, M.D., Ph.D., Study Chair — Chosun University Hospital
Locations (1):
- Chosun University Hospital, Gwangju, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koo CH, Ryu JH. Anesthetic considerations for urologic surgeries. Korean J Anesthesiol. 2020 Apr;73(2):92-102. doi: 10.4097/kja.19437. Epub 2019 Dec 17. PMID 31842248